CLINICAL TRIAL: NCT02629744
Title: A PHASE 1, OPEN-LABEL, SINGLE-ARM STUDY IN HEALTHY SUBJECTS TO EVALUATE PAIN, TOLERABILITY, SAFETY, AND USABILITY OF A PREFILLED AUTOINJECTOR TO SELF-ADMINISTER ETROLIZUMAB SUBCUTANEOUSLY
Brief Title: A Study to Evaluate Pain, Tolerability, Safety, and Usability of a Single Self-administered Etrolizumab by Auto-injector in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: GX29503
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — etrolizumab

ARMS (1):
- Etrolizumab (Experimental): Participants will self-administer single SC dose of etrolizumab using prefilled auto-injector, into the abdomen or the anterior thigh.
  Interventions: Drug: Etrolizumab; Device: Prefilled Auto-injector (Rotaject)

INTERVENTIONS:
Drug: Etrolizumab — Single SC dose of etrolizumab at 105 milligrams (mg) on Day 1.
  Other Names: rhuMAB Beta7
Device: Prefilled Auto-injector (Rotaject) — Participants self-administered etrolizumabSC injection using a prefilled auto-injector.

SUMMARY:
This study is a multi-center, single-arm, open-label study in healthy participants to assess the pain, tolerability, injection leakage, safety, and usability of a single self-administered subcutaneous (SC) dose of etrolizumab. Some participants will receive "needle-experience" training using a needle and syringe on Days -7 and -5, and health care professionals (HCPs) will then assess the participant's suitability to self-inject with a prefilled auto-injector (AI). The remainder of participants will be "needle naïve" and will not have previously self-injected. Eligible" needle experienced" and" needle naive" participants will attend an AI training visit at the study site on Day -3 (three days prior to etrolizumab dosing on Day 1). Following training and simulated injections by the participant the HCP will determine if the participant is suitable to proceed to actual etrolizumab dosing. All eligible study participants will self administer a single dose of etrolizumab (by AI) on Day 1 and will be followed up to Day 85 following dosing. Pain, tolerability, safety and usuability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, between 18 and 65 years of age, inclusive
* Within body mass index (BMI) range 18.0 to 32.0 kilograms per square meter (kg/m^2), inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead electrocardiograms (ECGs), and vital signs
* Females will be non-pregnant, non-lactating, and either postmenopausal (at least 1 year of non therapy induced amenorrhea), surgically sterile (absence of ovaries and/or uterus) for at least 90 days, or agree to remain abstinent or use a highly effective method of contraception for at least 24 weeks after the single dose of study drug
* Males will either be sterile or agree to remain abstinent or use a highly effective method of contraception for at least 24 weeks after the single dose of study drug. Male participants will refrain from sperm donation from Check-in (Day -1) until 24 weeks following study drug administration

Exclusion Criteria:

* Participation in any other investigational study drug or biological agent trial (including investigational vaccines) in which receipt of an investigational study drug occurred within 30 days or 5 half-lives or receipt of a biologic agent occurred within 90 days or 5 half-lives, whichever is longer, prior to Check-in (Day -1) and during the entire study
* Any prior treatment with etrolizumab or other anti integrin agents (including natalizumab, vedolizumab, and efalizumab)
* Any prior exposure to immunosuppressive agents (e.g., methotrexate, azathoprine, mercaptopurine)
* Use of IV steroids within 30 days prior to Screening;
* Chronic nonsteroidal anti inflammatory drug (NSAID)
* Use of any prescription medications/products within 14 days prior to Check in (Day -1)
* History of demyelinating disease
* Neurological conditions or diseases
* History of cancer
* History of alcoholism or drug addiction within 1 year prior to Check-in (Day -1)
* History of active or latent tuberculosis (TB), regardless of treatment history
* History of recurrent opportunistic infections, severe disseminated viral infections (e.g., herpes), or any serious opportunistic infection within the last 6 months
* Positive for human immunodeficiency virus (HIV) antibody
* Any current or recent signs or symptoms of infection
* Inability to sense pain (e.g., peripheral neuropathy) and have a history of or have been diagnosed with a chronic pain syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing Greater Than Mild Pain Immediately Following Injection at Time 0 Minute by 7-point Verbal Descriptive Scale (VDS-7) | 0 minute (immediately following injection)

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Greater Than Mild Pain Over Time by VDS-7 | 5, 10, 20, 60 minutes and 4 hours following injection
Percentage of Participants in each VDS-7 over time | 0 (immediately following injection), 5, 10, 20, 60 minutes, and 4 hours following injection
Mean Visual Analog Scale (VAS) over time | 0 (immediately following injection), 5, 10, 20, 60 minutes, and 4 hours following injection
Mean change from baseline in VAS over time | 0 (immediately following injection), 5, 10, 20, 60 minutes, and 4 hours following injection
Percentage of Participants With Injection-Site Reactions | 5 minute to Day 85 (end of study)
Percentage of Participants With Probable Root-causes of AI Usage Errors | Up to 4 hours following injection

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - Cypress, California
  - Dallas, Texas

REFERENCES:
- [Derived] Tyrrell H, Ravanello R, Pulley J, Tang MT, Zhang W, Abouhossein M, Tole S. An Open-Label Tolerability and Actual-Use Human Factors Study of Etrolizumab Autoinjector in Healthy Volunteers. Adv Ther. 2021 May;38(5):2406-2417. doi: 10.1007/s12325-021-01651-8. Epub 2021 Mar 29. PMID 33778928